CLINICAL TRIAL: NCT06882551
Title: Comparison of Intravitreal Bevacizumab Injection with Combination of Suprachoroidal Triamcinolone Acetonide Along with Intravitreal Bevacizumab Injection in the Treatment of Diabetic Macular Edema in Pseudophakic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Imran Ahmad, Assistant Professor Ophthalmology, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KhyberTeH; 450/DME/KMC (Other: Instititional Ethical and Review Board (IERB))
Record Dates: First submitted 2024-11-10; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Macular Edema (DME)
Keywords: intravitreal bevacizumab; suprachoroidal triamcinolone; diabetic macular edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravitreal Bevacizumab alone for center involving diabetic macular edema (Experimental): Effect of intravitreal Bevacizumab 1.25mg on center involving diabetic macular edema
  Interventions: Drug: Intravitreal Bevacizumab IVB
- Suprachoroidal triamcinolone acetonide and intravitreal Bevacizumab (Experimental): Combination of suprachoroidal triamcinolone acetonide and intravitreal Bevacizumab for the treatment of diabetic macular edema
  Interventions: Drug: intravitreal bevacizumab and suprachoroidal triamcinolone acetonide

INTERVENTIONS:
Drug: Intravitreal Bevacizumab IVB — Intravitreal bevacizumab alone
  Arms: Intravitreal Bevacizumab alone for center involving diabetic macular edema
Drug: intravitreal bevacizumab and suprachoroidal triamcinolone acetonide — Combination of Intravitreal bevacizumab and suprachoroidal triamcinolone acetonide
  Arms: Suprachoroidal triamcinolone acetonide and intravitreal Bevacizumab

SUMMARY:
Patients were included in the study who were pseudophakic with center-involved (sub-foveal) diabetic macular edema

DETAILED DESCRIPTION:
Patients were included in the study who were pseudophakic with center-involved (sub-foveal) diabetic macular edema. Those patients who had glaucoma history or IOP above 21 mm of Hg, Phakic, corneal opacity, vitreous hemorrhage, proliferative diabetic retinopathy, already received anti-VEGF injections, history of pan-retinal photocoagulation for proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with center involving diabetic macular edema on optical coherence tomography

Exclusion Criteria:

* Raised intraocular pressure
* History of glaucoma
* Corneal opacity
* Vitreous hemorrhage
* Proliferative diabetic retinopathy
* Anti-VEGF injections in last 3 months
* History of pan-retinal photocoagulation
* Contraindications for anti-VEGF

Ages: 32 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Central macular thickness | 3 months
  Effect of both treatment on central macular thickness measure on optical coherence tomography
Visual Acuity | 3 months
  Improvement in best corrected visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Teaching Hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Suprachoroidal injection of triamcinolone acetonide plus intravitreal bevacizumab in diabetic macular edema: a randomized pilot trial — https://pubmed.ncbi.nlm.nih.gov/36707790/